CLINICAL TRIAL: NCT00545844
Title: An 8 Week Study to Evaluate the Effectiveness of Adding Montelukast to Inhaled Corticosteroid (ICS) to the ICS/Long-Acting Beta 2-Agonist Therapy in Adult Subjects With Asthma and Allergic Rhinitis
Brief Title: Singulair(R) In Asthma And Allergic Rhinitis (0476-383)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0476-383; MK0476-383; 2007_024
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2009-08-19 (Estimated); Last update posted 2024-05-23 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

ARMS (1):
- 1 (Experimental): montelukast sodium
  Interventions: Drug: montelukast sodium

INTERVENTIONS:
Drug: montelukast sodium — montelukast sodium, 10 mg, one tablet once a day for 8 weeks as add on therapy to usual current asthma controller treatment
  Other Names: Singulair

SUMMARY:
Effectiveness of adding montelukast to inhaled corticosteroids in adult subjects with both uncontrolled asthma and allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a user of Inhaled Corticosteroid (ICS) or ICS/Long-Acting Beta 2-Agonist (ICS/LABA) at any dosage
* Peak expiratory flow is > or = 80% of predicted value on the day of visit 1
* Uncontrolled as per Canadian asthma consensus guidelines

Exclusion Criteria:

* Unwilling to stop regular use of histamine H1 antagonists for allergic rhinitis symptoms
* Unwilling to stop use of antihistamine eye drops or cromoglycate eye drops or ophthalmic corticosteroid

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2007-04-01 (Actual); Primary Completion 2008-01-01 (Actual); Study Completion 2008-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keith PK, Koch C, Djandji M, Bouchard J, Psaradellis E, Sampalis JS, Schellenberg RR, McIvor RA. Montelukast as add-on therapy with inhaled corticosteroids alone or inhaled corticosteroids and long-acting beta-2-agonists in the management of patients diagnosed with asthma and concurrent allergic rhinitis (the RADAR trial). Can Respir J. 2009 May-Jun;16 Suppl A(Suppl A):17A-31A. doi: 10.1155/2009/145071. PMID 19557208

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First 25 asthmatic patients seen consecutively at each site were invited to participate.
  Treatment phase: From the Survey population, blocks of 8 were allowed to participate. All subjects took 1 tablet of montelukast 10 mg once a day at bedtime.
  First patient in: APR-02-2007 Last patient out: JAN-25-2008
Pre-assignment Details: The anticipated Enrollment was 440, with an expected rate of 20% over the 8-week period, thus 369 patients should complete the study.
Groups:
- All Patients: montelukast sodium, 10 mg, one tablet once a day for 8 weeks as add on therapy to usual current asthma controller treatment
  Patients with comorbid allergic rhinitis and uncontrolled asthma were invited to participate in the treatment phase of the study. Of the 1004 patients who completed the survey phase, there were 319 eligible patients who advanced and participated in the treatment phase. Of the 319 eligible patients who advanced to the treatment phase 6 did not meet inclusion criteria leaving 313 patients.
Period: Overall Study
Arm/Group | All Patients
Started | 313
Completed | 301
Not Completed | 12
Not completed — Lost to Follow-up | 9
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 313
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199
  Male | 114
Inhaled Corticosteroids or Inhaled Corticosteroids / Long-Acting Beta 2-Agonist Use [Number; unit: participants]
  Inhaled Corticosteroids Only | 154
  Inhaled Corticosteroids/Long-Acting Beta 2-Agonist | 153
  Missing | 6
Allergic Rhinitis Diagnosis Duration [Mean (Standard Deviation); unit: Months] | 131.4 (135.4)
Asthma Diagnosis Duration [Mean (Standard Deviation); unit: Months] | 147.6 (139.0)

OUTCOME MEASURES:

1. Primary Outcome: Asthma Control
Description: Asthma control was assessed by the Canadian Asthma Consensus Guidelines at week 0 and week 8. Patients were considered uncontrolled if they answered "yes" to at least 2 of the 8 asthma control parameters.
Time Frame: 8 weeks (from Week 0 to Week 8)
Population: 319 patients advanced to the treatment phase and 313 patients qualified for inclusion in the intent to treat (ITT) analysis and completed the first visit. The following results are based on the 301 patients who completed week 8.
Measure: Number; unit: Participants
Arm/Group | Treatment Phase (All Patients) Week 0 | Treatment Phase (All Patients) Week 8
Number analyzed (Participants) | 313 | 301
Participants
  Uncontrolled | 312 | 72
  Controlled | 0 | 229
  Missing | 1 | 0

2. Secondary Outcome: The Mean Change in Mini Rhinoconjunctivitis Quality of Life Questionnaire (MiniRQLQ) Overall Score
Description: Mini Rhinoconjunctivitis Quality of Life Questionnaire (MiniRQLQ) consists of 14 questions to assess patient's overall quality of life related to allergic rhinitis on a scale of 0 (least impairment) to 6 (greatest impairment). The score is the mean of the 14 questions, ranging from 0 to 6. Change is computed as Week 8 score - Week 0 score
Time Frame: 8 weeks (from Week 0 to Week 8)
Population: Based on ITT population; there were 286 patients with available data regarding the mean change in MiniRQLQ at week 8.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Treatment Phase (All Patients) Week 8
Number analyzed (Participants) | 286
Units on a Scale | -1.45 (1.35)
Statistical Analysis 1: Comparison: Treatment Phase (All Patients) Week 8; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

3. Secondary Outcome: Effectiveness of Montelukast Therapy Used in Combination With Inhaled Corticosteroids or Inhaled Corticosteroids / Long-Acting Beta 2-Agonist in Improving the Symptoms of Asthma Using the Asthma Control Questionnaire (ACQ)
Description: The Asthma Control Questionnaire consists of 7 specific questions that were used to assess patient asthma control at week 0 and week 8. The mean score per question is used to determine the level of control, with a final score ranging from 0 (well-controlled) to 6 (extremely poorly controlled) units on a scale.
Time Frame: 8 weeks (from Week 0 to Week 8)
Population: There were 313 patients who qualified for inclusion in the intent to treat (ITT) analysis and completed the first visit; of these, 300 patients completed the ACQ at week 8.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Treatment Phase (All Patients) Week 0 | Treatment Phase (All Patients) Week 8
Number analyzed (Participants) | 313 | 300
Units on a Scale | 2.03 (0.80) | 0.92 (0.80)
Statistical Analysis 1: Comparison: Treatment Phase (All Patients) Week 0 vs Treatment Phase (All Patients) Week 8; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

4. Other Pre Specified Outcome: Patient Global Satisfaction
Description: At week 0 and week 8, patients were asked to complete a single question describing how satisfied they were regarding their asthma controller medication.
Time Frame: 8 weeks (from Week 0 to Week 8)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Treatment Phase (All Patients) Week 0 | Treatment Phase (All Patients) Week 8
Number analyzed (Participants) | 313 | 301
Participants
  Very satisfied | 24 | 136
  Satisfied | 77 | 110
  Neither satisfied or dissatisfied | 104 | 36
  Dissatisfied | 97 | 16
  Very dissatisfied | 11 | 1
  Missing | 0 | 2
Statistical Analysis 1: Comparison: Treatment Phase (All Patients) Week 0 vs Treatment Phase (All Patients) Week 8; McNemar-Bowker test is McNemar chi-squared statistic for binary matched pairs, with Bowker chi-squared fit test of symmetry model (tests all rows of data) (cf. Agresti, 2007); Test type: Superiority or Other; p < 0.001, McNemar-Bowker

5. Other Pre Specified Outcome: Physician Global Satisfaction
Description: At week 0 and week 8, physicians were asked to complete a single question describing how satisfied they were regarding their patient's asthma controller medication.
Time Frame: 8 weeks (from Week 0 to Week 8)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Treatment Phase (All Patients) Week 0 | Treatment Phase (All Patients) Week 8
Number analyzed (Participants) | 313 | 301
Participants
  Very satisfied | 7 | 135
  Satisfied | 54 | 110
  Neither satisfied or dissatisfied | 104 | 30
  Dissatisfied | 142 | 25
  Very dissatisfied | 4 | 1
  Missing | 2 | 0
Statistical Analysis 1: Comparison: Treatment Phase (All Patients) Week 0 vs Treatment Phase (All Patients) Week 8; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, McNemar-Bowker

6. Other Pre Specified Outcome: Patient Global Allergic Rhinitis Symptoms Assessment
Description: At week 0 and week 8, patients were asked to complete one question describing their perception of their allergic rhinitis symptoms.
Time Frame: 8 weeks (from Week 0 to Week 8)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Treatment Phase (All Patients) Week 0 | Treatment Phase (All Patients) Week 8
Number analyzed (Participants) | 313 | 301
Participants
  A non-issue as I do not have these symptoms | 11 | 41
  Not really bothersome | 35 | 129
  Bothersome a little of the time | 73 | 77
  Bothersome some of the time | 91 | 40
  Bothersome a good bit of the time | 94 | 13
  Missing | 9 | 1
Statistical Analysis 1: Comparison: Treatment Phase (All Patients) Week 0 vs Treatment Phase (All Patients) Week 8; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, McNemar-Bowker

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/313
Other Adverse Events (participants affected / at risk) | 11/313
OTHER ADVERSE EVENTS (reported when occurring in more than 0.3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=313)
Allergic reaction Not Otherwise Specified (Immune system disorders) | 1 (1)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma aggravated (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 1 (1)
Upset stomach (Gastrointestinal disorders) | 1 (1)
Muscular pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.